CLINICAL TRIAL: NCT05783765
Title: Role of Energy Balance Behaviors in Modifying Biobehavioral Risk Factors for Childhood Obesity
Brief Title: Food Genetics Behavior Study
Acronym: FOODIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 852728
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heightened Drive to Eat (Experimental): * Eating rate
  * Eating in the absence of hunger
  * Relative reinforcing value of food
  Interventions: Behavioral: Heightened Drive to Eat

INTERVENTIONS:
Behavioral: Heightened Drive to Eat — Participants' eating rate and eating in the absence of hunger will be assessed during a videotaped experimental meal. The relative reinforcing value of food will be assessed using a computerized behavioral choice task.

SUMMARY:
A genetic risk for obesity does not always translate to the development of obesity among children, which points to the presence of risk-modifying factors that likely relate to energy balance behaviors as key behavioral drivers. Using an integrated approach to comprehensively examine the interplay between genotype and phenotype, this study will systematically assess the extent to which energy balance behaviors, alone or in combination, in conjunction with family-level influences can modify behavioral and genetic predispositions to childhood obesity in a high-risk sample of predominantly minority children from low-resource backgrounds. Identifying protective factors that may mitigate the impact of obesity risk on weight and adiposity outcomes is critical for moving the prevention of childhood obesity into a new direction.

DETAILED DESCRIPTION:
This study examines the interplay between genotype and phenotype and assesses if energy balance behaviors in the context of the family environment, alone or in combination, can modify behavioral and genetic predispositions to childhood obesity. The research aims to prospectively evaluate the extent to which associations of a heightened drive to eat (HDE) on 1-year changes in weight and adiposity outcomes are independent or additive to those of a genetic risk for obesity among children. In addition, the study aims to prospectively examine risk-modifying energy balance behaviors in areas of diet, physical activity, and sleep that may mitigate the detrimental impact of a HDE or high genetic risk on weight and adiposity outcomes and test whether these factors differ for HDE versus a high genetic risk of obesity on those outcomes. Lastly, the research aims to examine the impact of family-level influences in areas of family functioning and parent feeding on risk-modifying energy balance behaviors in children.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* Children ages 5-7 years
* Children with BMI equal to or greater 5th percentile
* Mother must be children's biological mother and primary caregiver
* Mother must be able to read and understand English

Exclusion Criteria:

* Children with serious medical conditions or medication use known to affect food intake, body weight, physical activity, or sleep
* Children with developmental and/or psychiatric conditions that may impact study compliance
* Children with food allergies related to study foods or lactose intolerance
* Children with low preference for study foods

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 242 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Change from baseline to 1-year follow-up
  BMI z-score
Waist circumference | Change from baseline to 1-year follow-up
  Abdominal waist circumference (cm)
Body fat | Change from baseline to 1-year follow-up
  Body fat percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Penn Medicine Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No